CLINICAL TRIAL: NCT05332093
Title: Spatial Analysis of Host-parasite Interactions in the Skin Across the Clinical Spectrum of Cutaneous Leishmaniasis in Ethiopia
Brief Title: Spatial Analysis of Host-parasite Interactions in Cutaneous Leishmaniasis in Ethiopia
Acronym: SpatialCL
Status: Completed | Type: Observational
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: University of Gondar (Other); University of York (Other); Maastricht University (Other); University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Other Study IDs: 1451/20
Record Dates: First submitted 2022-03-08; First posted 2022-04-18 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Cutaneous Leishmaniases
Keywords: leishmania; leishmaniasis; cutaneous leishmaniasis; neglected tropical disease; immunoparasitology
MeSH Terms: conditions — Leishmaniasis, Cutaneous; Leishmaniasis; Neglected Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Blood, stool and skin samples will be isolated from CL patients and solely skin samples from healthy controls.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Local cutaneous leishmaniasis patients group (LCL): local cutaneous leishmaniasis patients
  Interventions: Diagnostic Test: skin biopsy; Diagnostic Test: venous blood sample (plasma, PBMC, WB); Genetic: venous blood sample (HLA); Genetic: skin slit
- Mucocutaneous leishmaniasis patients group (MCL): mucocutaneous leishmaniasis patients
  Interventions: Diagnostic Test: skin biopsy; Diagnostic Test: venous blood sample (plasma, PBMC, WB); Genetic: venous blood sample (HLA); Genetic: skin slit
- Diffuse cutaneous leishmaniasis patients group (DCL): diffuse cutaneous leishmaniasis patients
  Interventions: Diagnostic Test: skin biopsy; Diagnostic Test: venous blood sample (plasma, PBMC, WB); Genetic: venous blood sample (HLA); Genetic: skin slit
- Healthy control patients group Ethiopia (HC - Ethiopia): healthy control patients undergoing elective surgery in Northern Ethiopia
  Interventions: Diagnostic Test: skin biopsy
- Healthy control patients group Belgium (HC - Belgium): healthy control patients undergoing plastic surgery in Belgium
  Interventions: Diagnostic Test: skin biopsy

INTERVENTIONS:
Diagnostic Test: skin biopsy — 4mm skin biopsy
Diagnostic Test: venous blood sample (plasma, PBMC, WB) — venous blood sample to acquire plasma, PBMCs and whole blood
  Groups: Diffuse cutaneous leishmaniasis patients group (DCL); Local cutaneous leishmaniasis patients group (LCL); Mucocutaneous leishmaniasis patients group (MCL)
Genetic: venous blood sample (HLA) — venous blood sample used for HLA typing
  Groups: Diffuse cutaneous leishmaniasis patients group (DCL); Local cutaneous leishmaniasis patients group (LCL); Mucocutaneous leishmaniasis patients group (MCL)
Genetic: skin slit — genome sequencing of parasite DNA that is extracted from the skin slit
  Groups: Diffuse cutaneous leishmaniasis patients group (DCL); Local cutaneous leishmaniasis patients group (LCL); Mucocutaneous leishmaniasis patients group (MCL)

SUMMARY:
Cutaneous leishmaniasis manifestations range from self-healing localized skin ulcers/nodules to diffusely spread chronic lesions. Knowledge on the host-parasite interactions underpinning the different clinical presentations is scarce, in particular for L. aethiopica infections where disease can be extremely severe. Our aim is to define differences in skin immune responses and parasite virulence in CL patients at single cell/parasite level and how it underpins the different clinical presentations (localised, mucocutaneous and diffuse), by producing the first spatially-resolved 'ecological' map of the lesions.

DETAILED DESCRIPTION:
Specific objectives:

1. To profile the full heterogeneity in skin and lesion immunity (single cell RNAseq), and the cellular microenvironment surrounding infected and non-infected macrophages (digital spatial profiling).
2. To study the genomic diversity of L. aethiopica and identify features associated with the different clinical presentations (whole genome sequencing).
3. To understand how parasites respond to the microenvironmental conditions and define parasite survival niches (digital spatial profiling).
4. Study metabolic determinants of skin immunity (e.g. lipid metabolism, bioenergetics, short-chain fatty acids) in the context of key structural features of the skin landscape known to influence local metabolism and immune response (e.g. adipose tissue, follicles, microvasculature) (SpatialOMx).
5. To investigate the association between patient outcomes and the above host/parasite factors at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent
* Clinically confirmed CL diagnosis
* Between 12 and 50 years of age

Exclusion Criteria:

* Difficult or too painful sampling zone (see skin biopsy procedure below)
* (Primary) lesion size < 1 cm
* Already receiving CL treatment or received CL treatment in the last 3 months (excluding traditional medicine)
* Known major comorbidity at time of diagnosis (e.g. VL, HIV, TB, malaria, severe intestinal helminth infection)
* Medical history of VL
* Severely underweight (BMI<16)
* Known pregnancy
* Use of immunosuppressive medication in the last month
* Known excessive alcohol use (between >10 intakes/day and >10 intakes/week)
* History of hypersensitivity to local anaesthetics
* Presence of keloids/hypertrophic scars

Ages: 12 Years to 50 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients presenting at the LRTC and Boru Meda Hospital with clinically suspected CL during the study period will be screened for eligibility. Suspicion for CL is assessed by physicians as per routine care. In general, children are included in the study population since they are commonly affected, and also make up the majority of DCL patients.
Sampling Method: Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Spatially resolved immunological characterization of the CL lesion using single cell RNA sequencing and digital spatial profiling | Day 0
  Using single cell RNA sequencing and digital spatial profiling methods, we will profile the full heterogeneity in healthy skin/lesion immunity and the cellular microenvironment surrounding infected and non-infected macrophages, respectively.
Genomic characterization of L. aethiopica using whole genome sequencing | Day 0
  Whole genome sequencing will allow us to study the genomic diversity of L. aethiopica and identify features associated with the different clinical presentations.
Defining microenvironment and parasite niches in CL lesions using digital spatial profiling | Day 0
  The digital spatial profiling will indicate the different microenvironmental conditions and parasite survival niches.
Spatially resolved determination of the metabolic profile of the CL lesion using spatial OMx | Day 0
  The metabolic determinants of skin immunity (e.g. lipid metabolism, bioenergetics, short-chain fatty acids) in the context of key structural features of the skin landscape known to influence local metabolism and immune response (e.g. adipose tissue, follicles, microvasculature) will be studied by SpatialOMx.
The association between host/parasite factors and patients after treatment using clinical parameters | Month 6
  Patients are clinically assessed at day 0 (baseline visit), day 28 and month 6. These clinical assessments include a medical questionnaire and lesion assessment, and are compared with the single cell RNA sequencing and spatial resolution data to define potential causal relations between patient outcomes and immunometabolic factors.

CONTACTS AND LOCATIONS:
Overall Officials: Wim Adriaensen, PhD, Principal Investigator — Institute of Tropical Medicine Antwerp; Mikias Woldetensay, MD, Principal Investigator — University of Gondar
Locations (1):
- University of Gondar, Gonder, Amhara, Ethiopia

IPD SHARING:
Plan to Share IPD: Yes
IPD accessible by managed access
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After completion of the primary publication
Access Criteria: Applicants will need to fill out a data access request form
URL: https://www.itg.be/E/data-sharing-open-access